CLINICAL TRIAL: NCT02661555
Title: Effects of Aerobic Exercise on Brain Health in People With Multiple Sclerosis
Brief Title: Aerobic Exercise and Brain Health in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Jascha Fonden (Other); Knud and Edith Eriksens memorial fund (Unknown); University of Southern Denmark (Other); Augustinus fund (Unknown); Masku Neurological Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Brain health in MS
Record Dates: First submitted 2016-01-15; First posted 2016-01-22 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2018-05

CONDITIONS: Multiple Sclerosis; Brain Atrophy; Cognitive Impairment
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic exercise (Experimental): Aerobic exercise two times per week for 24 weeks.
  Interventions: Other: Aerobic exercise
- Habitual lifestyle (No Intervention): Habitual lifestyle the first 24 weeks. Will be offered the same exercise intervention after 24 weeks.

INTERVENTIONS:
Other: Aerobic exercise
  Arms: Aerobic exercise

SUMMARY:
The purpose of the project is to investigate how aerobic exercise affects brain volume, specific brain regions, neurotrophins and cognition in patients with multiple sclerosis.

The study will be a single blinded randomized controlled trial with a 6 months intervention.

It is hypothesized that aerobic exercise can slow down brain atrophy, increase the size of hippocampus, upregulate the secretion of neurotrophins and improve cognitive performance in people with multiple sclerosis.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a physically and cognitively disabling, chronic autoimmune disease of unknown etiology. It is the most common neurological disease affecting young adults in Western countries. According to the Danish MS Registry the prevalence has increased markedly over the last 40 years for particularly women, and today there are approximately 14.000 patients with MS (PwMS) in Denmark.

The pathological hallmark of MS is sclerotic plaque. Plaques in the central nervous system (CNS) can be detected in vivo using magnetic resonance imaging (MRI). Both the accumulation of lesions and the accelerated whole-brain atrophy correlate with the progressing physical and cognitive disabilities that clinically characterize PwMS.

The disease causes damage of both white and grey matter in the CNS, leading to whole brain atrophy and topographically specific atrophy within the hippocampus and the frontal and temporal cortices. The degradation of the CNS manifests as cognitive and physical disability. Cognitive impairment is estimated to affect up to 65% of PwMS, making it one of the most common and disabling symptoms of MS. Medical therapies for cognitive impairment in MS have so far proved ineffective. Collectively, the prevalence, impact and missing treatments highlight the importance of alternative approaches towards preservation of cognitive function. Despite equivocal findings, aerobic exercise represents a promising approach towards preservation or even expansion of hippocampal volume and cognitive functioning in MS. No longitudinal randomized controlled trial (RCT) study has so far applied the MRI technique when evaluating the potential neuro-protective effect of exercise on brain structure and function in MS. Also, given the scarcity of effective treatments for cognitive impairment in MS, a longitudinal exercise intervention evaluating the potential effect of aerobic exercise on cognition is urgently needed in MS.

The purpose of the present project is to investigate how aerobic exercise affects brain volume, specific brain regions, neurotrophins and cognition in PwMS.

It is hypothesized that aerobic exercise can slow down brain atrophy, increase the size of hippocampus, upregulate the secretion of neurotrophins and improve cognitive performance in people with MS.

The study will be a single blinded RCT. The exercise intervention will contain 6 months of aerobic training (bicycling, rowing and cross trainer) performed two times a week at moderate to high intensity and under supervision. The control group will be "living as usual" and will be offered the same exercise intervention after a 6 month period. A total of approximately 85 PwMS will be expected to be enrolled. The primary outcome of the study will be brain atrophy determined by MRI.

The current interdisciplinary project aims to document and understand the possible neuro-protective effects of exercise in MS. This would be of high relevance to PwMS (and other neurological pathologies). From a societal perspective it would help optimize MS rehabilitation and subsequently reduce MS related costs due to disability. In case of positive findings, this would provide the first convincing human evidence of a disease modifying effect of exercise in MS.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent
* Definite MS diagnosis
* Be clarified with the diagnosis and treatment
* Expectedly able to carry out the aerobic training / test
* Expanded Disability Status Scale (EDSS) score ≤6.0
* Must be able to transport themselves to and from training sessions

Exclusion Criteria:

* Dementia, alcohol abuse or pacemaker
* Medical comorbidity such as cardiovascular, respiratory, orthopedic or metabolic disorders or other concurrent diseases causing disability and hindering participation in the intervention
* Disease relapse in a 8 week period prior to study start
* Pregnancy
* Metallic implants hindering the MRI scans.
* Expected training attendance below 85%

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2016-01; Primary Completion 2018-08 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Percentage brain volume change | 0, 24 and 48 weeks

SECONDARY OUTCOMES:
Cognition measured by the Brief Repeatable Battery of Neuropsychological Tests | 0, 24 and 48 weeks
Blood samples: Cytokines and neurotrophins | 0, 24 and 48 weeks
  brain derived neurotrophic factor and key cytokines
VO2max | 0, 24 and 48 weeks
Regional volume change changes (e.g. hippocampus, thalamus) | 0, 24 and 48 weeks
Modified Fatigue Impact Scale | 0, 24 and 48 weeks
  Lower score is better. Range 0-84
Fatigue Severity Scale | 0, 24 and 48 weeks
  Lower score is better. Range 9-63.
Major Depression Inventory | 0, 24 and 48 weeks
  Lower score is better. Range 0-50
Short Form 36 | 0, 24 and 48 weeks
  Higher score is better. Each item is scored on a 0 to 100 range.
Multiple Sclerosis Impact Scale 29 | 0, 24 and 48 weeks
  Converted to a 0-100 scale where 100 indicates greater impact of disease on daily function
6-min walk test | 0, 24 and 48 weeks
  Walk as far as possible in 6 minutes. Higher is better.
Six Spot Step Test | 0, 24 and 48 weeks
  Complete the task as fast as possible. Faster is better.

CONTACTS AND LOCATIONS:
Overall Officials: Martin L Christensen, MSc, Principal Investigator — University of Aarhus
Locations (1):
- Sport Science, Department of Public Health, Aarhus University, Aarhus, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kupjetz M, Langeskov-Christensen M, Riemenschneider M, Inerle S, Ligges U, Gaemelke T, Patt N, Bansi J, Gonzenbach RR, Reuter M, Rosenberger F, Meyer T, McCann A, Ueland PM, Eskildsen SF, Nygaard MKE, Joisten N, Hvid L, Dalgas U, Zimmer P. Persons With Multiple Sclerosis Reveal Distinct Kynurenine Pathway Metabolite Patterns: A Multinational Cross-Sectional Study. Neurol Neuroimmunol Neuroinflamm. 2025 Nov;12(6):e200461. doi: 10.1212/NXI.0000000000200461. Epub 2025 Sep 18. PMID 40966534
- [Derived] Langeskov-Christensen M, Grondahl Hvid L, Nygaard MKE, Ringgaard S, Jensen HB, Nielsen HH, Petersen T, Stenager E, Eskildsen SF, Dalgas U. Efficacy of High-Intensity Aerobic Exercise on Brain MRI Measures in Multiple Sclerosis. Neurology. 2021 Jan 12;96(2):e203-e213. doi: 10.1212/WNL.0000000000011241. Epub 2020 Dec 1. PMID 33262230
- [Derived] Langeskov-Christensen M, Hvid LG, Jensen HB, Nielsen HH, Petersen T, Stenager E, Hamalainen P, Dalgas U. Efficacy of high-intensity aerobic exercise on cognitive performance in people with multiple sclerosis: A randomized controlled trial. Mult Scler. 2021 Sep;27(10):1585-1596. doi: 10.1177/1352458520973619. Epub 2020 Nov 24. PMID 33232191